CLINICAL TRIAL: NCT05048420
Title: THE EFFECT OF RAMP LESION REPAIR ON RETURN TO SPORTS IN ANTERIOR CRUCIATE LIGAMENT RECONSTRUCTION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Emre DANSUK, lecturer, Medipol University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: MedipolUni
Record Dates: First submitted 2021-09-01; First posted 2021-09-17 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: ACL; Meniscus Lesion; Sport Injury
Keywords: ramp lesion; acl; return to sport
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ramp lesion repair (Experimental)
  Interventions: Procedure: surgery
- Anterior cruriciate ligament reconstruction (Experimental)
  Interventions: Procedure: surgery

INTERVENTIONS:
Procedure: surgery — ACL reconstruction and RAMP lesion repair

SUMMARY:
Purpose/reason of the research: The anterior cruciate ligament (ACL) is an important ligament in maintaining knee function. In patients with anterior cruciate ligament (ACL) injury, concomitant intra-articular lesions are usually seen. It has been reported that approximately 43% of all patients with ACL tears have associated lateral or medial meniscal injuries.

Injury associated with a tear of the meniscotibial ligament in the posterior horn of the medial meniscus is defined as a RAMP lesion. Because the RAMP lesion is located within the posteromedial "blind spot", it has historically been underdiagnosed.

It has been reported that 9-17% of all ACL tears have RAMP lesions. RAMP lesions have been found to increase the force on the ACL. Injury to the meniscotibial ligaments has been shown to increase rotational instability of the knee.

Based on the available literature, there is a discrepancy between authors regarding the repair of a RAMP lesion during an acute ACL surgery. In chronic ACL rupture, some authors have suggested that the RAMP lesion has a suitable biological environment for healing.

thinks. However, excessive mobility of the meniscocapsular junction has been reported in RAMP lesions during knee flexion and extension. It has been suggested that these lesions are different from other peripheral tears and are not suitable for spontaneous healing. It is suggested that meniscal RAMP lesion repair will be the most effective approach. Rehabilitation after repair of a RAMP lesion depends on whether the repair is performed concurrently with ACL surgery. When performed with an ACL surgery, the process is followed according to the ACL rehabilitation protocol.

Even if the functionality of the knee is fully restored in the post-ACL surgery period, not all patients can return to their previous level of sportive performance due to various psychological, social and physiological factors. In the literature, different information can be found as criteria for returning to sports after ACL surgery. The rate of returning to sports was reported as 65-88% in patients with ACL reconstruction, and 19-82% in patients who were followed conservatively. However, there are few studies with short- or long-term follow-up after the identification and treatment of RAMP lesions. Accordingly, our aim in this study is to comprehensively evaluate the return to sports of participants who have undergone isolated anterior cruciate ligament surgery and who have had simultaneous RAMP lesion repair with anterior cruciate ligament surgery.

This assessment will provide the opportunity to examine functional capacity, balance, psychological state, activity level and pain with different measurement methods.

Material and method of the research: The study will consist of 2 groups, including 12 participants who have undergone isolated ACL surgery and 12 participants who have had simultaneous RAMP lesion repair in Istanbul Medipol Mega Hospitals Complex Orthopedics and Traumatology Unit, with a total of 24 participants.

ELIGIBILITY:
Inclusion Criteria:

* ACLR
* ACLR with RAMP lesion repair
* To complete the 9th month after surgery
* Home exercise program by physiotherapist after surgery

Exclusion Criteria:

* Additional pathologies requiring surgery other than anterior cruciate ligament and RAMP lesion
* Misalignment
* Other ligamentous lesions
* Cartilage pathologies
* Joint disorders
* History of surgery from the same knee
* Chronic inflammatory and rheumatological disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Return to Sports After Anterior Cruciate Ligament Injury Scale (ACL-RSI) | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided